CLINICAL TRIAL: NCT05393115
Title: Does Inspiratory Pressure Wave Form Influence Respiratory Muscle Fatigue and Metabolism During Resistive Breathing
Brief Title: Respiratory Muscle Fatigue at Different Breathing Modes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Mathias Krogh Poulsen, Teaching Associate Professor, Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Eso_pres_fatigue
Record Dates: First submitted 2022-04-21; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Square wave breathing — difference in time to failure from the two breathing modes
  Other Names: Triangle wave breathing

SUMMARY:
The study aims at investigating if time to respiratory muscle fatigue and metabolism are influenced by the pressure wave form mode applied during resistive breathing.

DETAILED DESCRIPTION:
In healthy subjects fitted with a nasogastric double balloon catheter and breathing at a resistance, the investigators will measure time to failure, Borg ratings, VO2, VCO2, flow, esophageal-, gastric- and airway-pressure. This will be done during breathing at either a square wave or triangle wave pressure waveform, in random order and trials separated by >two days. Further respiratory muscle fatigue will be investigated pre and post intervention by maximal esophageal pressure generation (voluntary and with cervical magnetic stimulation).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women
* Age ≥18 and ≤60 years
* BMI ≥ 20 and ≤30

Exclusion Criteria:

* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous and present neurologic (e.g. ataxia), musculoskeletal (e.g. muscular dystrophy) or mental illnesses (e.g. schizophrenia)
* History of mechanical ventilation, COVID-19 with respiratory complications, lung cancer
* Part of lung resected
* Presence of dyspepsia/heart-burn/abdominal pain
* Presence of esophageal varices
* Presence of liver disease
* Presence of esophageal hernia
* Pregnancy
* Failure to comply with transcranial magnetic stimulation adult safety screen
* History of epilepsy, metal implants in head or jaw
* Acute or chronic lung diseases, e.g. asthma, COPD, bronchitis etc.
* Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to task failure (Tlim) | Up to two months between the two different breathing trials (randomized order)
  The time (s) from the subject starts to breathe under the experimental condition, and until task failure will be measured. Task failure is defied by either subject intolerance to continue or by lacking ability of the subject to maintain the target pressure and/or timing. From a previous publication (Bellemare and Grassino, JAP, 1982), it is estimated that subjects will reach Tlim between 30min to 1 hour. If breathing is continued after 1 hour, task failure will not happen as breathing can be continued indefinitely.

SECONDARY OUTCOMES:
Respiratory muscle pressures | Up to two months between the two different breathing trials (randomized order)
  Respiratory muscle pressure will be measured by esophageal and gastric pressure (in cmH2O) using a naso gastric catheter fitted with double balloons (Nutrivent) connected to a pressure sensor (ICU lab, KleisTek).
Tidal volume | Up to two months between the two different breathing trials (randomized order)
  Tidal Volume (ml) will be measured with a flowsensor (Hans Rudolph) through a pressure box (ICU lab, KleisTek)
Respiratory work | Up to two months between the two different breathing trials (randomized order)
  Work of breathing (j), will be calculated from outcome measure 2 and 9 (pressure (cmH2O) and insp. and expiratory time (s)). Measured with pressure box (ICU lab, KleisTek)
Ratings of perceived exertion | Up to two months between the two different breathing trials (randomized order)
  Borg Dyspnea Scale, from 0-10 where 0 is no effort at all and 10 is maximal breathing effort.
Metabolism | Up to two months between the two different breathing trials (randomized order)
  Energy expenditure calculated from VO2 (ml/min) nad VCO2 (ml/min) with e.g Weir equation. VO2 and VCO2 are measured with Beacon (Mermaid care).
Respiratory rate | Up to two months between the two different breathing trials (randomized order)
  Respiratory rate (breaths/min) will be measured with a flowsensor (Hans Rudolph) through a pressure box (ICU lab, KleisTek)
Minute ventilation | Up to two months between the two different breathing trials (randomized order)
  Minyte ventilation (l/min) will be measured with a flowsensor (Hans Rudolph) through a pressure box (ICU lab, KleisTek)
Insp. and expiratory time | Up to two months between the two different breathing trials (randomized order)
  Insp. and expiratory time (s) will be measured with a flowsensor (Hans Rudolph) through a pressure box (ICU lab, KleisTek)

CONTACTS AND LOCATIONS:
Locations (1):
- Mathias Krogh Poulsen, Aalborg, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No